CLINICAL TRIAL: NCT05924854
Title: The Influence of Electroacupuncture on Postoperative Agitation of Sevoflurane Inhalation Combined With Intravenous Anesthesia in Pediatrics: an Experimental, Single-center Clinical Study
Brief Title: The Influence of Electroacupuncture on Postoperative Agitation of Pediatrics Undergoing Sevoflurane General Anesthesia
Acronym: DZDXEQFWQMSHZD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Leihuajuan, Principal Investigator, The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019XJJJ040
Record Dates: First submitted 2023-05-30; First posted 2023-06-29 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: General Anesthetics Toxicity; Postoperative Cognitive Dysfunction; Electroacupuncture
Keywords: Electroacupuncture; Sevoflurane; Postoperative agitation; pediatrics
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: Randomization according to center will be used. Subjects were randomly assigned to the sevoflurane general anesthesia group（S group） and the electroacupuncture group（E group） at a ratio of 1:1.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Due to the particularity of acupuncture research, acupuncturist only carries out electroacupuncture. Blinded evaluation visitor will be used in the trial, and the efficacy will be evaluated by a third party not envovled in assignments. Blind statistical analysis was used in the data summary stage, and the researchers, operators and statisticians were separated to ensure the authenticity and reliability of the study results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (E group) (Experimental): When the patient's vital signs are stable, the blind researcher (acupuncturist) checks the electroacupuncture device, (SDZ-Ⅱ, Suzhou Medical Supplies Factory),after the check is been done, acupuncturist uses Huatuo brand copper milli-needle needles to pierce Baihui point（DU20）, Shenting point (DU24), bilateral Zulinqi (GB41) and bilateral Taichong (LR3) , and fixed and connection them to SDZ-Ⅱ..At first, sets the device output to zero ,then .the acupuncturist turns on the power of the treatment instrument with the output frequency from 50 to 100hz on a weak to strong wave mode continuously , 20 min after the intervention, stops the machine, the acupuncturist turns off the device and pulls out the needles.
  Interventions: Other: electroacupuncture
- sevoflurane general anesthesia group（S group） (No Intervention): Anesthesia induction, anesthesia maintenance and anesthesia monitoring will carry out exactly the same in both groups,only difference is that S group has no electroacupuncture intervention.

INTERVENTIONS:
Other: electroacupuncture — Electroacupuncture (EA) is a method of treating diseases by inserting a needle (usually a filiform needle) into the skin or tissue of a patient at a certain Angle, and then passing through the needle (sensing) micro-current waves of human bioelectricity to stimulate specific parts of the human body (acupoints). Equipment used in the trial included:
  1. Huatuo brand copper filiform needle (diameter: 0.35×50mm), Suzhou Medical Supplies Factory, Food and Drug Administration firearms production: Suzhou Food and Drug Administration firearms production No. 20010020.
  2. Electroacupuncture apparatus: SDZ-Ⅱ electroacupuncture apparatus of Huatuo brand, Suzhou Medical Supplies Factory Co., LTD., Registration No. : 20172270675
  Arms: Electroacupuncture group (E group)

SUMMARY:
Postoperative agitation is a common complication in pediatric anesthesia, with an incidence ranging from 10% to 80%. Common surgical procedures in children include tonsillectomy, adenoidectomy, insidious penis prolongation and circumcision, etc. Postoperative delirium and agitation is a clinical emergency, and can have detrimental effects on the child's health. The primary clinical manifestations include disorganized movements, moaning, incoherent speech, confusion and paranoid characters, inability to be concentrated, and irritability, obstinacy or uncooperative; all these would increase the risks of falling out of bed, possible fractures, and all kinds of tube loss. These symptoms would sustain postoperative recovery significantly and pose a possible long-term neurological dysfunction. As a result, an extended hospitalization, elevated in-hospital mortality rate, escalated medical expenses, heightened risk of cognitive impairment, reduced quality of life, and increased incidence of postoperative complications.

Traditional acupuncture has been shown to improve cerebral micro-circulation, correct energy metabolism disorders, alleviate chronic pain and regulate visceral function, lessen fatigue and modulate immune. Moreover, acupuncture is a simple, effective and safe therapy. Electroacupuncture therapy is produced and developed on the basis of acupuncture therapy, which has a regulatory effect on multiple systems of the body and can play a regulatory effect that is consistent with normal physiological regulation. Modern medicine believes that the anterior cingulate gyrus, hippocampus, and other regions of the limbic system are the possible center control of emotion and cognition. Electroacupuncture treatment can help accelerate the recovery of central nervous system function, which plays a protective role on the central nerve system, especially the brain, within 24-72 hours after electroacupuncture treatment. At the same time, electroacupuncture is beneficial to the recovery of immune function postoperatively, it can promote the release of central neurotransmitters and improve receptor activity, so as to play a role in postoperative analgesia, reduce the dosage of anesthetics, brain protection, neurological function rehabilitation, and so on. According to scientific research, it also posses a certain effect on the prevention and treatment of postoperative delirium. Sevoflurane is an inhale anesthetic which is widely used in clinics for pediatric general anesthesia. Due to the high incidence of postoperative delirium and agitation, it has been given rise to great concern on pediatric clinical anesthesia. In order to reduce delirium and agitation incidence, the investigators apply electroacupuncture in pediatric for sevoflurane combined with intravenous general anesthesia, aim to target a safe way to lessen postoperative brain complications on pediatric.

This is a single-center experimental study that employs randomization, triple-blinding, and control study. Pediatric patients were randomly assigned to two groups, sevoflurane general anesthesia group (S group) and electroacupuncture group (E group), 40 patients, respectively. Anesthesia induction, maintenance, and monitoring be performed identically in both groups, the S group will not receive electroacupuncture treatment, the E group will receive electroacupuncture therapy. Electroacupuncture intervention will be performed by blinded acupuncture physicians, visitor who is blind to collect preoperative, intraoperative and postoperative data while visiting patients, data statisticians, who are blind to the intervention, data collection, conducted statistical analyses on the data electronically.

DETAILED DESCRIPTION:
Pediatric patients who meet the screening criteria were randomly divided into two groups,sevoflurane general anesthesia group (S group) and electroacupuncture group (E group), 40 patients in each group, respectively. Anesthesia induction, maintenance, and monitoring performed identically in both groups, the S group will not receive electroacupuncture treatment, the E group will receive electroacupuncture therapy. All patients have a regular preoperative fasting, monitoring of vital signs after the patient was admitted to the operating room, Preoxygenation was performed by face mask oxygen with oxygen flow set to 8 L/min for 3 minutes to each patient, and anesthesia induced with 8% sevoflurane inhalation while oxygen flow rate will set to 2 L/min. After the patient slept and accessing successful venipuncture, intravenous drugs were administered with midazoline 0.03-0.05 mg/kg, propofol 0.3-0.5 mg/kg, sufentanil 0.4-0. 5 mg/ kg, and cisatracurium 0.15 mg/kg for induction of anesthesia. After the patient's muscle relaxation, tracheal intubation was performed, and the patient's airway pressure was monitored by connecting an airway pressure detection device, and then IPPV-controlled ventilation was performed by connecting a Drager Fabius GS anesthesia machine (Drager Germany), with oxygen flow rate set to 1 L/min, initial tidal volume set to 6-8 ml/kg, and initial respiratory rate set to 15-20 bpm, adjusted to PaCO2 was maintained at about 36-40 mmHg. The patient's depth of anesthesia was also detected with the EEG dual frequency index, and the BIS was about 45-50.

After general anesthesia induction, the acupuncturist used a Huatuo brand copper milli-needle (Suzhou Medical Supplies Factory) and selected Baihui point（DU20）, Shenting point (DU24), bilateral Zulinqi (GB41) and bilateral Taichong (LR3) point, for acupuncture. The acupuncture points are located 5 inches straight up from the middle of the front hairline of the head, and 0.3-0.5 inches from the midpoint of the front and back hairline of the patient's head in a 1-inch deviation. The TaiChong (LR3) point is located on the back of the patient's foot between the 1st and 2nd metatarsal bones, in the depression in front of the union of the metatarsal bones, or when the patient's foot artery is pulsating, the point is taken from the patient's 1st and 2nd metatarsal bones and pushed backward to the bottom, with a vertical puncture of 0.5-0.8 inch; the foot Linobu (GB41) point is located on the back of the patient's foot, in front of the union of the 4th and 5th metatarsal bones, on the outside of the 5th toe extensor tendon, with a vertical stab of 0.3-0.5 inch.

Then,the acupuncturist check the EA device ( SDZ-Ⅱ,Suzhou Medical Supplies Factory)before use, the EA device is set to zero at the beginning, then connect the acupuncture needle to the EA device and fixed, output frequency of EA from weak to strong (50-100hz) ,use sparse and dense mode,after 20 minutes intervention, pause the EA output, turn off the electric power ,and pulled out the needle. all the acupoint pressed by the Cotton swabs until there is no bleeding.

Maintenance of anesthesia: Patients were given continuous intraoperative inhalation of 1% sevoflurane combined with continuous intravenous propofol 5 mg.kg-1h-1 sevoflurane inhalation will be discontinued 30 minutes before the end of surgery, and propofol was stopped immediately after surgery. The inhalation concentration of sevoflurane adjusting according to the depth of anesthesia, intermittent intraoperative injection of sufentanil and cisatracurium, and other anesthetic drugs stopped at the end of surgery. All the pediatric anesthesia will be carried out by the anesthesiologists. Intraoperative BP, HR, MAP, RR, SpO2, infusion fluid and bleeding volume, total anesthetic dosage all keep record in time by the anesthesiologists. The anesthesia depth measures by Bispro (BeliveA2) and maintains between 40-60.

All patients are transferred to the PACU at the end of surgery, the patient's ECG, HR, MAP, RR, and SpO2 are monitored all the time. The tracheal tube is removed after the patient was fully awake, and recovery and extubation time keeps in record, PAED scale, Wong-bank facial expression scale, Ramsay sedation score recorded, adverse events of anesthesia like nausea, and vomiting all recorded 2 hours, 24 hours, 72 hours postoperatively; as well as anal exhaust time and defecate time. Venous blood sampling for inflammatory factors is carried out preoperative, 24 hours and 72 hours postoperatively.

In this experiment, the blinded investigator (acupuncturist) will perform the electroacupuncture intervention on the patients, the blinded investigator (assess visitor) will collect the data, and the blinded data statistician will analyze the data by computer and perform the statistical analysis. It will be performed using SPSS 17.0 statistical analysis software. All statistical tests were performed using a two-sided test, and a p-value less than or equal to 0.05 was considered a statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

1. Age 4-13 years old, both sexes;
2. Tonsillectomy, adenoidectomy, concealed penis, and circumcision were planned under sevoflurane intravenous inhalation combined general anesthesia;
3. The weight of the children was 10-60kg;
4. The child had no history of allergy or mental disease.
5. No respiratory tract infection within two weeks;
6. No infection at the puncture site;
7. There was no significant difference in body weight, age and operation time between the electroacupuncture group (E group) and the sevoflurane general anesthesia group（S group）.
8. The informed consent was signed by the legal guardian of the patient before surgery.

Exclusion Criteria:

1. Age < 4 years old, age > 13 years old;
2. Body weight < 10kg, body weight > 60kg;
3. The child has a history of heart disease, asthma, mental disease, and major surgery;
4. A history of respiratory infection in the past two weeks;
5. Non-electroacupuncture indications;
6. Infection at the acupuncture site;
7. Patients with liver and kidney insufficiency, cardiopulmonary insufficiency;
8. Those with allergic constitution (allergic to two or more substances);
9. Persons with legal disabilities;
10. Refusal to sign the consent form;

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Pediatric Anesthesia Emergence Delirium Scale | 24 hours before surgery,
  PAED is one of the commonly used scales in clinical practice. The scale includes 5 items, and the scores of each item are summed to obtain the PAED score. The higher the score, the more severe the degree of delirium.
Pediatric Anesthesia Emergence Delirium Scale | 2 hours after extubation in PACU
  PAED is one of the commonly used scales in clinical practice. The scale includes 5 items, and the scores of each item are summed to obtain the PAED score. The higher the score, the more severe the degree of delirium.
Pediatric Anesthesia Emergence Delirium Scale | 24 hours after surgery
  PAED is one of the commonly used scales in clinical practice. The scale includes 5 items, and the scores of each item are summed to obtain the PAED score. The higher the score, the more severe the degree of delirium.
Pediatric Anesthesia Emergence Delirium Scale | 72 hours after surgery
  PAED is one of the commonly used scales in clinical practice. The scale includes 5 items, and the scores of each item are summed to obtain the PAED score. The higher the score, the more severe the degree of delirium.

SECONDARY OUTCOMES:
Wong-bank(FPS-R) | 24 hours before surgery, 2 hours after extubation in PACU, and 24 hours and 72 hours after surgery.
  FPS-R asks participants to rate their global pain level on a scale of 0 (no pain) to 10 (worst pain). Fp- R provides cartoon images of six facial expressions (ranging from smiling to sad to painful crying) to represent the pain level. For the assessment, the patient points to a scale or cartoon face that corresponds to his or her pain level
visual analogue scale (VAS) | 24 hours before surgery, 2 hours after extubation in PACU, and 24 hours and 72 hours after surgery
  Visual analogue Scale (VAS) is the most commonly used single-dimensional measurement of pain intensity. The scale mainly consists of a 10-cm straight line, one end of which indicates "no pain at all" and the other end indicates "the most severe pain imaginable" or "pain to the extreme" etc. The patient is asked to mark the corresponding position on the line (with a dot or a "✕" etc.) to indicate the intensity of the pain they feel at the time.
Inflammatory markers in venous blood | 24 hours before surgery, 2 hours after extubation in PACU, and 24 hours and 72 hours after surgery.
  The following indexes were observed: IL-6, IL-8, CPR, S-100β, NSE, SOD, TNF-α.
Sequencing analysis of the gut microbiota | 24 hours before surgery, 2 hours after extubation in PACU, and 24 hours and 72 hours after surgery.
  The human gut is home to a large number of microorganisms, also a place for absorption, energy metabolism, immune regulation, and many disease.By observing the time of nausea, vomiting, anal exhaust and defecation (and collecting feces)time,, This is the first time to explore whehter gut flora plays an important role on peadatric agitation postoperatively. The study of intestinal flora is of great significance on peadatric agitation undergoing sevoflurane general anesthesia with the electroacupuncture intervention .

OTHER OUTCOMES:
The wake recovery time of the patient after the operation | the patient is transfer to the pacu and observe 2 hours after the extubation.
  The wake recovery time of the patient after the operation (the patient is transfer to the pacu and observe 2 hours after the extubation ).

CONTACTS AND LOCATIONS:
Overall Officials: Feng Zhong, Doctor, Principal Investigator — Hunan University of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Hunan University of Chinese Medicine, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Describe the IPD sharing plan, including what IPD are to be shared with other researchers：